CLINICAL TRIAL: NCT00977405
Title: Collagen-Gentamicin Implant in the Treatment of Contaminated Surgical Abdominal Wounds - A Randomized Controlled Trial
Brief Title: Collagen-Gentamicin Implant in the Treatment of Contaminated Surgical Abdominal Wounds
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Novem Healthcare Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Collatamp G
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Superficial Surgical Site Infection
Keywords: Wound infection; Gentamicin; Contaminated wounds
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Primary closure after standard washing of wound with chlorhexidine solution
- Collatamp G (Experimental): Primary closure of wound with collatamp G in subcutaneous layer
  Interventions: Device: Collatamp Gentamicin Implant

INTERVENTIONS:
Device: Collatamp Gentamicin Implant — Collatamp Gentamicin placed into subcutaneous layer of dirty abdominal wounds
  Other Names: CollatampG
  Arms: Collatamp G

SUMMARY:
The investigators' hypothesis is that placement of CollatampG in the subcutaneous layer of contaminated abdominal wounds is effective prophylaxis for superficial surgical site infection (SSI). CollatampG is composed of highly purified type 1 collagen obtained from bovine tendon, which acts as a vehicle for the aminoglycoside antibiotic, gentamicin. This implant provides a high concentration of local gentamicin at the surgical wound to decrease the local microorganism load. It has been shown that if a surgical site is contaminated with > 10 to the power of 5 microorganisms per gram of tissue, the risk of infection is markedly increased. When a gastrointestinal organ is the source of pathogens, gram-negative bacilli (e.g., E. coli) are typical isolates, which are susceptible to gentamicin. Therefore, a high local concentration of gentamicin at the contaminated surgical wound provided by the CollatampG implant may prevent the local bacterial load from reaching levels high enough to cause a clinical infection.

DETAILED DESCRIPTION:
Aims: To decrease the incidence of superficial surgical site infection (SSI) using a collagen -gentamicin implant (CollatampG) for patients who undergo major abdominal surgery with contaminated surgical wounds.

Hypotheses: Patients undergoing abdominal surgery with wounds classified as contaminated or dirty are at a high risk of SSI. Wounds are classified as contaminated when an operation is performed through an infected area (e.g abscess, perforated viscus or traumatic wound) that has been exposed for over 4 hours. Risk of infection in these wounds has been shown to be as high as 45 %.

Our hypothesis is that placement of CollatampG in the subcutaneous layer of contaminated abdominal wounds is effective prophylaxis for superficial SSI. CollatampG is composed of highly purified type 1 collagen obtained from bovine tendon, which acts as a vehicle for the aminoglycoside antibiotic, gentamicin. This implant provides a high concentration of local gentamicin at the surgical wound to decrease the local microorganism load. It has been shown that if a surgical site is contaminated with >10 to the power of 5 microorganisms per gram of tissue, the risk of infection is markedly increased. When a gastrointestinal organ is the source of pathogens, gram-negative bacilli (e.g., E. coli) are typical isolates, which are susceptible to gentamicin. Therefore, a high local concentration of gentamicin at the contaminated surgical wound provided by the CollatampG implant may prevent the local bacterial load from reaching levels high enough to cause a clinical infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a preoperative diagnosis of perforated viscus, perforated gastrointestinal tumour, or intraabdominal abscess (based on clinical and radiological findings), requiring abdominal surgery.
* Patient with prolonged surgery (operative time charted > 4 hours).
* Age 21 and above, able to understand the information regarding the study.
* Agreeable for randomization and signed consent form.

Exclusion Criteria:

* Patients who have known allergy to products of bovine origin or to the antibiotic, gentamicin.
* Pregnant women or breast-feeding mothers.
* No signed consent form.
* Intra-operative surgical finding inconsistent with inclusion criteria (lack of evidence of intra-peritoneal sepsis or duration of surgery < 4 hours).
* Patients having urgent abdominal surgery without indication of intra-peritoneal sepsis (such as patients with impending intestinal obstruction).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of superficial surgical site infections | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Julian KP Ong, FRCSEd, Principal Investigator — Singapore General Hospital; Jit-Fong Lim, FRCS, Study Director — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Guzman Valdivia Gomez G, Guerrero TS, Lluck MC, Delgado FJ. Effectiveness of collagen-gentamicin implant for treatment of "dirty" abdominal wounds. World J Surg. 1999 Feb;23(2):123-6; discussion 126-7. doi: 10.1007/pl00013171. PMID 9880419
- [Result] Poulsen KB, Bremmelgaard A, Sorensen AI, Raahave D, Petersen JV. Estimated costs of postoperative wound infections. A case-control study of marginal hospital and social security costs. Epidemiol Infect. 1994 Oct;113(2):283-95. doi: 10.1017/s0950268800051712. PMID 7925666